CLINICAL TRIAL: NCT00228514
Title: Sub Study: Controlled Rosuvastatin Multinational Study in Heart Failure (CORONA) PET Sub Study
Brief Title: Dutch Sub Study: Controlled Rosuvastatin Multinational Study in Heart Failure (CORONA). PET Sub Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4522IL/0098 Dutch SubStudy; D3562C00098
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2010-11

CONDITIONS: Rosuvastatin; Heart Failure; Positron Emission Tomography (PET)
MeSH Terms: conditions — Heart Failure | interventions — Rosuvastatin Calcium; Magnetic Resonance Spectroscopy

INTERVENTIONS:
Drug: Rosuvastatin
  Other Names: Crestor
Procedure: Positron emission tomography

SUMMARY:
At one site, patients participating in the Corona main study are asked to participate in the PET-substudy. Before and 6 months after study medication is started a Positron Emission Tomography (PET-scan) is performed to study the effect of rosuvastatin in Chronic Heart Failure on myocardial perfusion (reserve)

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling the in and exclusion criteria of the CORONA study and separate informed consent for participation in the sub study.

Exclusion Criteria:

* See above

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-02; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To study the effect of rosuvastatin in Chronic Heart Failure on myocardial perfusion (reserve). Before and 6 months after study medication is started a Positron Emission Tomography (PET-scan) is performed.

SECONDARY OUTCOMES:
To study the effect of rosuvastatin in Chronic Heart Failure on mismatch. Before and 6 months after study medication is started a Positron Emission Tomography (PET-scan) is performed.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca CV Medical Department, Study Director — AstraZeneca
Locations (1):
- Research Site, Groningen, Netherlands